CLINICAL TRIAL: NCT03568487
Title: Scapula Adaption in Overhead Athletes: Novel Scapulometer Development, Scapula Movement Adaption and Intensive Scapula-focused Intervention
Brief Title: Scapula Adaption in Overhead Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201712089RINC
Record Dates: First submitted 2018-05-30; First posted 2018-06-26 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-05

CONDITIONS: Scapular Dyskinesis
Keywords: scapular dyskinesis; EMG biofeedback; scapulometer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive scapula-focused approach (Experimental)
  Interventions: Other: Intensive scapula-focused approach
- Control therapy (Active Comparator)
  Interventions: Other: Control Therapy

INTERVENTIONS:
Other: Intensive scapula-focused approach — scapula-focused approach with exercises, 3 x 20 min training per week for 4 weeks
  Arms: Intensive scapula-focused approach
Other: Control Therapy — not have any physical training but is encouraged to stay active as usual.
  Arms: Control therapy

SUMMARY:
Previous studies have proposed various ways to assess scapular dyskinesis, but they were impractical in clinical setting or the validity was questioned. The novel scapulometer we developed can measure the prominence of scapular medial border and inferior angle. We would like to examine its reliability and validity in subjects with symptomatic scapular dyskinesis. The long-term, high-intensity, unilateral loading may cause overhead athletes to develop adaptive changes in shoulder kinematics, range of motion (ROM) and strength in the dominant arm. We hypothesized that these changes may be related to scapular dyskinesis. According to the previous studies, we expect electromyography (EMG) biofeedback training can help improve the ratio of muscle activation of scapular muscle.

DETAILED DESCRIPTION:
Fifty subjects of scapular dyskinesis will be classified and recruited from overhead players (baseball, basketball, tennis, volleyball, and so on) at high schools and through local Internet media. All participants and their legal guardians will provide written informed assent and consent, respectively, and the study will be approved by the Ethics Committee Institutional Review Board. Since intervention may be specific to pattern of scapular dyskinesis, pattern of scapular dyskinesis in control group will match the pattern of scapular dyskinesis in the intervention group. Twenty-five subjects per group is based on a minimal revenant difference of a self-reported functional questionnaire between intervention and control (Struyf et al., 2013; Andersen et al., 2014). Participants will be recognized as elite players in their age categories. Subjects will be excluded if they have a history of shoulder pain or injury. Players will supply their player characteristics, including years of sports practice, weekly sports and conditioning exposure and type of sports. Players' standing height, sitting height, and body mass will be measured and used with the chronologic age to estimate their biological age according to the assessments of skeletal age, dental age, and secondary sex characteristics (Baxter et al., 2005). A clinical trial with a blinded assessor will be conducted. The subject takes a form (with a letter A or B) indicating allocation to either groups (scapula-focused approach versus control) from a closed envelop. For the scapula-approached group, pattern of scapular dyskinesis will be assessed. Then subjects in B control group will meet pattern-matched criteria related to pattern assessment of scapula-focused group. More subjects may be recruited for the control group to meet pattern-matched criteria of scapula-approached group. A list with subject numbers and the group allocation that results from this matched-control procedure will be stored in a sealed envelope. Only the therapist has direct access to the allocation list. In this way, subjects are allocated to either intervention or control group comprised of 25 subjects in each group. Both groups will be treated by the same therapist.

ELIGIBILITY:
Inclusion Criteria:

* (1) with scapular dyskinesis
* (2) overhead players (baseball, basketball, tennis, volleyball, and so on) at high schools

Exclusion Criteria:

* if they have a history of shoulder pain or injury

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 170 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change of range of motion after 4-week training | Baseline and after 4-week training
  Passive interior rotation ROM and exterior rotation ROM of the glenohumeral joint will be assessed bilaterally using a hand-held standard universal goniometer. The player will lay supine with the humerus abducted to 90 degrees and elbow flexed to 90 degrees. The fulcrum of the goniometer is set at the olecranon process.
Change of muscle strength after 4-week training | Baseline and after 4-week training
  The maximal isometric strength of 8 shoulder-scapula complex muscles will be assessed bilaterally using a handheld dynamometer. Each test will be performed twice, with a 30-second rest period between tests. The largest strength value for each muscle will be used for statistical analyses, normalized to body weight (in kilograms), and expressed as a percentage for inter individual comparison.
Change of shoulder complex kinematics after 4-week training | Baseline and after 4-week training
  The Polhemus 3Space FASTRAK system (Polhemus Inc., Colchester, VT, USA) will be used to record shoulder complex kinematics.
Change of muscular activities after 4-week training | Baseline and after 4-week training
  Bipolar surface electromyographic (EMG) electrodes will be placed over the upper trapezius (UT), middle trapezius (MT), lower trapezius (LT), and serratus anterior (SA) of the dominant shoulder to record muscular activities.

SECONDARY OUTCOMES:
Forward shoulder posture (acromial distance) | Baseline and after 4-week training
  The measurement of the distance between the posterior border of the acromion and the table (acromial distance) is performed in supine. In this position, the assessor measured the distance between the most posterior aspect of the posterior border of the acromion and the table bilaterally.
Pectoralis minor muscle length | Baseline and after 4-week training
  The distance from the fourth rib to the coracoids process will be measured with FASTRAK system with accuracy of 0.08 cm. This distance (in centimeter) is divided by the subjects height and multiplied by 100. This results in a pectoralis muscle length index (PMI).

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, Taipei, Taiwan